CLINICAL TRIAL: NCT06590233
Title: The Risk Factors and Predictors of Hyperglycemia Secondary to Acute Pancreatitis
Brief Title: Hyperglycemia and Acute Pancreatitis
Status: Completed | Type: Observational
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Tuo Li, MD, Deputy Director, Shanghai Changzheng Hospital
Other Study IDs: NMU-3cDM-1A
Record Dates: First submitted 2024-08-29; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Acute Pancreatitis (AP); Diabetes Mellitus
Keywords: Acute pancreatitis; Diabetes mellitus; PPDM-A; Risk factor
MeSH Terms: conditions — Pancreatitis; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Acute pancreatitis

SUMMARY:
The goal of this observational study is to learn about post-acute pancreatitis diabetes mellitus (PPDM-A). The main questions it aims to answer are:

1. What are the clinical characteristics of PPDM-A?
2. What are the related factors for PPDM-A?

All patients with acute pancreatitis have been given standardized treatment for the condition.

The researchers will compare the PPDM-A group with the non-PPDM-A group to find the risk factors for PPDM-A.

DETAILED DESCRIPTION:
Investigators retrospectively collected data from patients with acute pancreatitis (AP) in participating centers between January 2013 and June 2024.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pancreatitis attending participating centers since January 2013 (patients with clinically reported AP (ICD-10:K85 or related diagnosis));
2. Age between 18 and 80 years;
3. Patients have undergone glucose metabolic tests at least 1 month after discharge from hospital.

Exclusion Criteria:

1. Patients with a history of diabetes mellitus prior to the AP attack;
2. Patients who underwent pancreatic surgery;
3. Patients with hereditary pancreatitis and autoimmune pancreatitis;
4. Patients with missing data regarding age or gender.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We collected data from patients with acute pancreatitis (AP) in participating centers between January 2013 and June 2024.
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2024-08 (Actual); Study Completion 2024-08 (Actual)

PRIMARY OUTCOMES:
Number of participants who have developed PPDM-A | From the AP treatment to 5 years after the end of treatment
  PPDM-A was defined as diabetes after AP in the absence of a history of preexisting diabetes before the AP episode.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bharmal SH, Cho J, Ko J, Petrov MS. Glucose variability during the early course of acute pancreatitis predicts two-year probability of new-onset diabetes: A prospective longitudinal cohort study. United European Gastroenterol J. 2022 Mar;10(2):179-189. doi: 10.1002/ueg2.12190. Epub 2022 Feb 20. PMID 35188346
- [Background] Bharmal SH, Cho J, Alarcon Ramos GC, Ko J, Stuart CE, Modesto AE, Singh RG, Petrov MS. Trajectories of glycaemia following acute pancreatitis: a prospective longitudinal cohort study with 24 months follow-up. J Gastroenterol. 2020 Aug;55(8):775-788. doi: 10.1007/s00535-020-01682-y. Epub 2020 Jun 3. PMID 32494905
- [Background] Zhong S, Du Q, Liu N, Chen Y, Yang T, Qin S, Jiang Y, Huang X. Developing a CT-based radiomics nomogram for predicting post-acute pancreatitis diabetes mellitus incidence. Br J Radiol. 2023 Dec;96(1152):20230382. doi: 10.1259/bjr.20230382. Epub 2023 Oct 24. PMID 37750855
- [Background] Lv Y, Zhang J, Yang T, Sun J, Hou J, Chen Z, Yu X, Yuan X, Lu X, Xie T, Yu T, Su X, Liu G, Zhang C, Li L. Non-Alcoholic Fatty Liver Disease (NAFLD) Is an Independent Risk Factor for Developing New-Onset Diabetes After Acute Pancreatitis: A Multicenter Retrospective Cohort Study in Chinese Population. Front Endocrinol (Lausanne). 2022 May 25;13:903731. doi: 10.3389/fendo.2022.903731. eCollection 2022. PMID 35692404
- [Background] Yu BJ, Li NS, He WH, He C, Wan JH, Zhu Y, Lu NH. Pancreatic necrosis and severity are independent risk factors for pancreatic endocrine insufficiency after acute pancreatitis: A long-term follow-up study. World J Gastroenterol. 2020 Jun 21;26(23):3260-3270. doi: 10.3748/wjg.v26.i23.3260. PMID 32684740
- [Background] Zhi M, Zhu X, Lugea A, Waldron RT, Pandol SJ, Li L. Incidence of New Onset Diabetes Mellitus Secondary to Acute Pancreatitis: A Systematic Review and Meta-Analysis. Front Physiol. 2019 May 31;10:637. doi: 10.3389/fphys.2019.00637. eCollection 2019. PMID 31231233
- [Background] Das SL, Singh PP, Phillips AR, Murphy R, Windsor JA, Petrov MS. Newly diagnosed diabetes mellitus after acute pancreatitis: a systematic review and meta-analysis. Gut. 2014 May;63(5):818-31. doi: 10.1136/gutjnl-2013-305062. Epub 2013 Aug 8. PMID 23929695
- [Background] Shen HN, Yang CC, Chang YH, Lu CL, Li CY. Risk of Diabetes Mellitus after First-Attack Acute Pancreatitis: A National Population-Based Study. Am J Gastroenterol. 2015 Dec;110(12):1698-706. doi: 10.1038/ajg.2015.356. Epub 2015 Nov 3. PMID 26526084